CLINICAL TRIAL: NCT01361932
Title: Speak Fast, Use Jargon, and Don't Repeat Yourself: Using Online Videos to Supplement Emergency Department Discharge Instructions
Brief Title: Using Online Videos to Supplement Emergency Department Discharge Instructions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Clare Atzema, MD MSc, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: AFP-CA-01
Record Dates: First submitted 2011-05-25; First posted 2011-05-27 (Estimated); Last update posted 2013-03-27 (Estimated); Status verified 2013-03

CONDITIONS: Emergency Department Discharge Instructions; Instruction Videos

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Video of ED Discharge Instructions (Experimental)
  Interventions: Other: Video of ED discharge instructions for patient's ED discharge diagnosis
- Control (usual standard of care) (No Intervention)

INTERVENTIONS:
Other: Video of ED discharge instructions for patient's ED discharge diagnosis — Link provided for a website of 38 ED discharge instruction videos, based on ED discharge diagnosis; patients in study group encouraged to view it upon returning home. Three key questions asked by RA 1 to 5 days later, via phone call, and answers scored.
  Arms: Video of ED Discharge Instructions

SUMMARY:
This project will evaluate the effectiveness of 38 videos of discharge instructions for patients seen in, and discharged from, the emergency department (ED). The investigators will (1) assess how many ED patients chose view the website, and (2) interview patients who viewed a video, as well as those who didn't view a video (and therefore received standard care), to determine whether patients who viewed a video understood their diagnoses and discharge instructions better.

ELIGIBILITY:
Inclusion Criteria:

* Age > 16, or < 16 and accompanied by a legal guardian
* Has one of 38 ED discharge diagnoses
* Fluent in English, or caregiver fluent
* Has access to a computer, with internet access, in the next 4 days
* Has access to a telephone

Exclusion Criteria:

* Age < 16 when unaccompanied by a legal guardian
* Decreased level of consciousness at ED discharge (eg palliative patient)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2011-11; Primary Completion 2012-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Score out of 3 points on 3 key questions | 1 to 5 days after ED visit
  3 key questions have been created for each of 38 ED discharge diagnosis. Scores will be compared between intervention group and control group.

SECONDARY OUTCOMES:
Quality rating of video of discharge instructions, Likert scale 1 to 5 | 1 to 5 days after ED discharge
  Rating by study arm (who viewed a video) as to how helpful the video was in helping them (1) understand their discharge instructions, and (2) overall usefulness of the video.

CONTACTS AND LOCATIONS:
Overall Officials: Clare L Atzema, MD MSc FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre

REFERENCES:
- [Derived] Atzema CL, Austin PC, Wu L, Brzozowski M, Feldman MJ, McDonnell M, Mazurik L. Speak fast, use jargon, and don't repeat yourself: a randomized trial assessing the effectiveness of online videos to supplement emergency department discharge instructions. PLoS One. 2013 Nov 11;8(11):e77057. doi: 10.1371/journal.pone.0077057. eCollection 2013. PMID 24244272